CLINICAL TRIAL: NCT07309731
Title: Impact OF Cooled Versus Thermal Radiofrequency Denervation In Management Of Chronic Lumber Facet Joint Pain.Prospective Study.
Brief Title: Impact OF Cooled Versus Thermal Radiofrequency Denervation In Management Of Chronic Lumber Facet Joint Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, manal mohamed rashad, lecturer, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1788/2-Nov-2025
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Lumber Facet Joint Pain(Lower Back Pain ) Relief by Cooled Radiofrequency or Thermal Radiofrequency Denervation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thermal radio frequency denervation (T) group (Active Comparator): The medial branch of the dorsal spinal ramus is the main target .The fluoroscopy will be then placed at slightly oblique view . An 22-gauge insulated RF needle with 1 cm active tip will be used .the parameters of Radiofrequency Denervation treatment are : the tip temperature being at 80 °C, 45V (volt), the frequency 2 Hz for 120 s, three cycles with rotation of the needle each time. At the end of the radiofrequency(RF)procedure, after the probe is removed , 20 mg methylprednisolone acetate will be given through the RF needle for each level
  Interventions: Device: thermal radio frequency denervation
- Cooled Radiofrequency denervation (C) group (Active Comparator): Patients will positioned prone with a C-arm fluoroscopy. 22-gauge spinal needles were placed in the appropriate location as lumbar medial branch blocks in Spinal Intervention Society Guidelines . 17-gauge 4 mm active tipped CRFA electrodes were used for the procedure . The CRFA (cooled radio frequency ablation) electrodes were also placed in the appropriate location similar to described as lumbar medial branch blocks procedure, instead of traditional placement of electrodes described as in Spinal Intervention Society Guidelines.The RFA generator temperature set to 60°C (intralesional temperature >80°) for 150 seconds for each
  Interventions: Device: Cooled Radiofrequency denervation

INTERVENTIONS:
Device: thermal radio frequency denervation — The medial branch of the dorsal spinal ramus is the main target .The fluoroscopy will be then placed at slightly oblique view . An 22-gauge insulated RF needle with 1 cm active tip will be used .the parameters of Radiofrequency Denervation treatment are : the tip temperature being at 80 °C, 45V, the frequency 2 Hz for 120 s, three cycles with rotation of the needle each time. At the end of the RF procedure, after the probe is removed , 20 mg methylprednisolone acetate will be given through the RF needle for each level
  Arms: thermal radio frequency denervation (T) group
Device: Cooled Radiofrequency denervation — Patients will positioned prone with a C-arm fluoroscopy. 22-gauge spinal needles were placed in the appropriate location as lumbar medial branch blocks in Spinal Intervention Society Guidelines . 17-gauge 4 mm active tipped CRFA electrodes were used for the procedure . The CRFA electrodes were also placed in the appropriate location similar to described as lumbar medial branch blocks procedure, instead of traditional placement of electrodes described as in Spinal Intervention Society Guidelines.The RFA (radio frequency ablation) generator temperature set to 60°C (intralesional temperature >80°) for 150 seconds for each
  Arms: Cooled Radiofrequency denervation (C) group

SUMMARY:
Chronic lumber facet joint pain is defined according to international association of study of pain (IASP)as multifactorial phenomenon of pain that persist more than 3 months after an injury and /or beyond the usual course of an acute lumber facet pain or a reasonable time for a comparable injury to heal .

lumber facet joint degeneration (LRFJ) is the 1st source of chronic low back pain with an incidence of 15% t o 45 % among patients with low back pain . the spinal facet joint has an abundant nerve supply ; therefore, pain can be caused by arthritic change, degenerative change, inflammation, and injury .

Degeneration of all LFJs (lumbar facet joints) was diagnosed using magnetic resonance image (MRI) , the most sensitive and diagnostic tool. Thus, hypertrophy, degeneration, and the accumulation of fluid within the joints are signs of LFJ degeneration it was found in all treated LFJs .

facet joint pain management can be achieved using medical therapy or facet joint therapeutic interventions, ultrasound guided injection,or fluoroscopically guided facet joint injection (FJI) , medial branch block (MBB) , or radiofrequency ablation .

Radiofrequency is a minimally invasive procedure and is operated under light

intravenous sedation or local anesthesia when necessary. Radiofrequency

energy is delivered to the target nerves through an insulated needle , and this

energy heats and denatures the nerve for the purpose of pain relief . The

radiofrequency techniques include, thermal, and cooled radiofrequency .

thermal radiofrequency (TRFA) uses more energy and higher temperature compared

with cooled radiofrequency , cooled radiofrequency ablation (CRFA) is a

newer technique, and may have some theoretical advantages over traditional

radiofrequency whereas , cooled radiofrequency adopts internally probes to

increase lesion size , and it can increase the chance of complete denervation .

based on heat neurotomy (60°C (celsius) vs. 80°C in TRFA) with the resulting ablative area twice as long and extending distally from the tip of the electrode.

ELIGIBILITY:
Inclusion Criteria:

* Patient's acceptance .
* Both sexes (male and female).
* Age between 30 and 70 years .
* Physical status; ASA I , II. (American society of anesthesiologist)
* BMI; 22-30 Kg/m2.
* Presence of

  1. Chronic Lumbar Facet Joint Pain (numerical rating scale (NRS) ≥ 6) lasting for 3 months or more without any response to noninvasive conservative treatment methods like NSAIDs and gabapentin therapy for pain control, or physiotherapy,
  2. Patients have two to three levels of bilateral facet arthropathy with normal motor power of lower extremities
  3. Local paraspinal tenderness with increased pain on hyperextension, rotation, or lateral bending of the lower lumbar spine.
* More than or equal to 50% temporary pain relief following an ultrasound guided diagnostic medial branch block with local anesthetic corticosteroid injection.

Exclusion Criteria:

* Those with spondylolisthesis or disc herniation or internal disc disruption (IDD).
* Previous spinal surgery at the level to be treated , Spinal canal stenosis or spinal instability.
* Patient with previous radiofrequency ablation.
* Patients having radicular pain, neurogenic claudication, or neurological deficits.
* Coagulopathy, bleeding disorders .
* Allergy to medications or contrast to be used .
* Rheumatic disorders.
* Systemic infections, or local infections in the field of intervention .
* Any uncontrolled medical or psychiatric condition .
* Pregnancy, lactating women .

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | NRS will be detected and recorded immediately 2 hours post intervention and then at 1 week , 1 month , 3 months, and 6 months after intervention .
  using a numerical rating scale (NRS) ranging from 0 to 10 (0: "no pain" to 10: "the worse pain")

CONTACTS AND LOCATIONS:
Overall Officials: khadeja m elhossieny, MD, Principal Investigator — Zagazig University
Locations (1):
- Faculty of Medicine,Zagazig University, Zagazig, Elsharqya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planed after completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: planed after completion of the study and publication
Access Criteria: principal investigator

REFERENCES:
- [Background] Cohen SP, Kapural L, Kohan L, Li S, Hurley RW, Vallejo R, Eshraghi Y, Dinakar P, Durbhakula S, Beall DP, Desai MJ, Reece D, Christiansen S, Chang MH, Carinci AJ, DePalma M. Cooled radiofrequency ablation versus standard medical management for chronic sacroiliac joint pain: a multicenter, randomized comparative effectiveness study. Reg Anesth Pain Med. 2024 Mar 4;49(3):184-191. doi: 10.1136/rapm-2023-104568. PMID 37407279
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Candan B, Gungor S. Cooled-radiofrequency neurotomy for the treatment of chronic lumbar facet (zygapophyseal) joint pain: A retrospective study. Medicine (Baltimore). 2021 Dec 30;100(52):e28459. doi: 10.1097/MD.0000000000028459. PMID 34967387
- [Background] Coluzzi F, Polati E, Freo U, Grilli M. Tapentadol: an effective option for the treatment of back pain. J Pain Res. 2019 May 16;12:1521-1528. doi: 10.2147/JPR.S190176. eCollection 2019. PMID 31190963
- [Background] Davidson M, Keating J. Oswestry Disability Questionnaire (ODQ). Aust J Physiother. 2005;51(4):270. doi: 10.1016/s0004-9514(05)70016-7. No abstract available. PMID 16358452
- [Background] Dunlevy C, MacLellan GA, O'Malley E, Blake C, Breen C, Gaynor K, Wallace N, Yoder R, Casey D, Mehegan J, Fullen BM, O'Shea D. Does changing weight change pain? Retrospective data analysis from a national multidisciplinary weight management service. Eur J Pain. 2019 Sep;23(8):1403-1415. doi: 10.1002/ejp.1397. Epub 2019 May 21. PMID 30963658
- [Background] Kwak DG, Kwak SG, Lee AY, Chang MC. Outcome of intra-articular lumbar facet joint corticosteroid injection according to the severity of facet joint arthritis. Exp Ther Med. 2019 Nov;18(5):4132-4136. doi: 10.3892/etm.2019.8031. Epub 2019 Sep 20. PMID 31616521
- [Background] Li SJ, Zhang SL, Feng D. A comparison of pulsed radiofrequency and radiofrequency denervation for lumbar facet joint pain. J Orthop Surg Res. 2023 May 5;18(1):331. doi: 10.1186/s13018-023-03814-5. PMID 37143095
- [Background] Manchikanti L, Kaye AD, Soin A, Albers SL, Beall D, Latchaw R, Sanapati MR, Shah S, Atluri S, Abd-Elsayed A, Abdi S, Aydin S, Bakshi S, Boswell MV, Buenaventura R, Cabaret J, Calodney AK, Candido KD, Christo PJ, Cintron L, Diwan S, Gharibo C, Grider J, Gupta M, Haney B, Harned ME, Helm Ii S, Jameson J, Jha S, Kaye AM, Knezevic NN, Kosanovic R, Manchikanti MV, Navani A, Racz G, Pampati V, Pasupuleti R, Philip C, Rajput K, Sehgal N, Sudarshan G, Vanaparthy R, Wargo BW, Hirsch JA. Comprehensive Evidence-Based Guidelines for Facet Joint Interventions in the Management of Chronic Spinal Pain: American Society of Interventional Pain Physicians (ASIPP) Guidelines Facet Joint Interventions 2020 Guidelines. Pain Physician. 2020 May;23(3S):S1-S127. PMID 32503359
- [Background] McCormick ZL, Choi H, Reddy R, Syed RH, Bhave M, Kendall MC, Khan D, Nagpal G, Teramoto M, Walega DR. Randomized prospective trial of cooled versus traditional radiofrequency ablation of the medial branch nerves for the treatment of lumbar facet joint pain. Reg Anesth Pain Med. 2019 Mar;44(3):389-397. doi: 10.1136/rapm-2018-000035. PMID 30777903
- [Background] Mukherjee K, Das A, Basunia SR, Dutta S, Mandal P, Mukherjee A. Evaluation of Magnesium as an adjuvant in Ropivacaine-induced supraclavicular brachial plexus block: A prospective, double-blinded randomized controlled study. J Res Pharm Pract. 2014 Oct;3(4):123-9. doi: 10.4103/2279-042X.145387. PMID 25535620
- [Background] Rubinstein SM, de Zoete A, van Middelkoop M, Assendelft WJJ, de Boer MR, van Tulder MW. Benefits and harms of spinal manipulative therapy for the treatment of chronic low back pain: systematic review and meta-analysis of randomised controlled trials. BMJ. 2019 Mar 13;364:l689. doi: 10.1136/bmj.l689. PMID 30867144
- [Background] Shih CL, Shen PC, Lu CC, Liu ZM, Tien YC, Huang PJ, Chou SH. A comparison of efficacy among different radiofrequency ablation techniques for the treatment of lumbar facet joint and sacroiliac joint pain: A systematic review and meta-analysis. Clin Neurol Neurosurg. 2020 Aug;195:105854. doi: 10.1016/j.clineuro.2020.105854. Epub 2020 Apr 19. PMID 32353665